CLINICAL TRIAL: NCT06572553
Title: Evaluation of Therapeutic Efficacy of Faricimab for Clinical AMD, DME, and RVO Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0612
Record Dates: First submitted 2024-08-13; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-03

CONDITIONS: Age-Related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
Keywords: Age-Related Macular Degeneration; Faricimab; Diabetic Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion | interventions — faricimab

STUDY DESIGN:
Intervention Model Description: 1. Chinese patients aged 18 years or older ;
  2. Patients who have been diagnosed with nAMD, DME or RVO by OCT, FFA, ICGA or OCTA;
  3. Patients whose decision to receive treatment with faricimab was made prior to and independent of study participation;
  4. Patients who have received at least one treatment with faricimab during the course of the study;
  5. have signed an informed consent form.
Masking Description: All roles know what drug they injected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of faricimab (Experimental): Intervention: Intravitreal Injections Generic name: faricimab Dosage: 0.05ml (6mg) Frequency: every month Duration: 3 months
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Faricimab (faricimab-svoa; Vabysmo), a bispecific antibody that inhibits both VEGF-A and Ang-2, was developed by Roche/Genentech, and dual-pathway inhibition may provide stronger and longer-lasting efficacy in the treatment of retinal vascular disease relative to anti-VEGF therapy alone.

SUMMARY:
The goal of this clinical trial is to learn if drug Faricimab works to treat nAMD, DME or RVO in adults. It will also learn about the safety of drug Faricimab. The main questions it aims to answer are:

Does drug Faricimab can improve the best-corrected visual acuity of participants? What medical problems do participants have when inject drug Faricimab? Participants will inject drug Faricimab every month for 3 months. Visit the clinic once every 2 weeks for checkups.

DETAILED DESCRIPTION:
Intravitreal anti-vascular endothelial growth factor (VEGF) therapies are used to treat retinal vascular diseases such as neovascular (wet) age-related macular degeneration (nAMD), diabetic macular edema (DME), and retinal vein occlusion (RVO). However, the clinical effectiveness of such therapies is often suboptimal, often resulting in poor treatment adherence due to the burden of frequent monitoring and injection therapy (every 4-8 weeks). Different approaches have been investigated to improve outcomes in such diseases, including modification of dosing regimens to reduce treatment burden and continued research to identify new drug targets. Angiopoietin-2 (Ang-2) has been implicated in the pathogenesis of several retinal vascular diseases, including nAMD and DME, and has therefore been identified as a potential new target.

Faricimab (faricimab-svoa; Vabysmo), a bispecific antibody that inhibits both VEGF-A and Ang-2, was developed by Roche/Genentech. Dual-pathway inhibition may provide stronger and longer-lasting efficacy in the treatment of retinal vascular disease. Faricimab is administered via intravitreal injection. It is the first bispecific antibody designed for intraocular use. In January 2022, faricimab was approved in the United States for the treatment of participants with nAMD or DME. And in March 2024, faricimab began to be approved for use in the treatment of patients in our clinic.

Therefore, investigators collected participants who were injected with Faricimab in the clinic and conducted follow-up visits to evaluate the therapeutic efficacy and application prospect of Faricimab in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese patients aged 18 years or older and of any gender;
2. Patients who have been diagnosed with nAMD, DME or RVO by OCT, FFA, ICGA or OCTA;
3. Patients whose decision to receive treatment with faricimab was made prior to and independent of study participation;
4. Patients who have received at least one treatment with faricimab during the course of the study;
5. have signed an informed consent form.

Exclusion Criteria:

1. Active ocular inflammation or suspected active ocular infection in either eye;
2. Receipt of any other anti-VEGF therapy after faricimab;
3. Patient is unable to provide clinical data (visual acuity and OCT images) within 2 weeks (14 days) prior to receiving the initial faricimab injection;
4. Currently participating in any other clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | through study completion, an average of 3 months.
  BCVA will be measured at a standard distance of 4 metres under standardised lighting conditions (85-100 candela) by using an ETDRS optometer. Each eye will be tested separately with the participants who wear best corrected vision glasses. The smallest line of letters that the patient can correctly identify will be recorded as their BCVA.Measurements will be taken by trained ophthalmologists at baseline and at time points such as 2 weeks after the start of the trial and 1 month after the start of the trial to ensure consistency.

SECONDARY OUTCOMES:
central retinal thickness (CRT) | through study completion, an average of 3 months.
  Retinal thickness will be measured by using optical coherence tomography (OCT). Patients will undergo standardised retinal imaging, performed after pupil dilation. The average retinal thickness in and around the central sulcus will be measured using an automatically generated thickness map from the OCT device.
Choroidal neovascularization (CNV) | through study completion, an average of 3 months.
  Choroidal neovascularisation was measured by OCT and OCTA. Standardised retinal imaging was performed after pupil dilation. Using the images provided by the OCT and OCTA devices, the presence or absence of accompanying choroidal neovascularisation was measured, and if present, the type was further determined

CONTACTS AND LOCATIONS:
Overall Officials: Panpan Ye, doctor, Study Director — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Basic characteristics,multimodal imaging data

REFERENCES:
- [Background] Ferro Desideri L, Traverso CE, Nicolo M, Munk MR. Faricimab for the Treatment of Diabetic Macular Edema and Neovascular Age-Related Macular Degeneration. Pharmaceutics. 2023 May 5;15(5):1413. doi: 10.3390/pharmaceutics15051413. PMID 37242655
- [Background] Stanga PE, Valentin-Bravo FJ, Stanga SEF, Reinstein UI, Pastor-Idoate S, Downes SM. Faricimab in neovascular AMD: first report of real-world outcomes in an independent retina clinic. Eye (Lond). 2023 Oct;37(15):3282-3289. doi: 10.1038/s41433-023-02505-z. Epub 2023 Mar 23. PMID 36959312
- [Background] Giancipoli E, Guglielmi A, Bux AV, Clima GME, Pignatelli F, Boscia F, Viggiano P, Boscia G, Fortunato F, Besozzi G, Niro A, Dore S, Iaculli C. Real-World Outcomes of a Loading Phase with Intravitreal Faricimab in Neovascular Age-Related Macular Degeneration (n-AMD) and Diabetic Macular Edema (DME). Ophthalmol Ther. 2024 Aug;13(8):2163-2184. doi: 10.1007/s40123-024-00980-5. Epub 2024 Jun 4. PMID 38831127